CLINICAL TRIAL: NCT02901821
Title: Predicting Concussion Outcomes With Salivary miRNA
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Steven Hicks, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: STUDY00003729
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary nucleic acids
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: No intervention. Collection of medical/demographic info and salivary RNA in children 5-21 years without history of mild traumatic brain injury (mTBI).
  Interventions: Genetic: salivary RNA collection
- Concussion: Collection of medical/demographic info and salivary RNA in children 5-21 years with history of mild traumatic brain injury (mTBI). Collection of PCSI concussion assessment interview tool and balance/cognition testing at time of injury, 1-2wks post injury, and 4wks post injury.
  Interventions: Genetic: salivary RNA collection

INTERVENTIONS:
Genetic: salivary RNA collection — collection of saliva for microRNA (small noncoding RNA) processing

SUMMARY:
The purpose of this study is to identify changes in salivary ribosomal nucleic acid (RNA) expression that are predictive of symptom duration and character following mild traumatic brain injury (mTBI) in children.

DETAILED DESCRIPTION:
The purpose of this study is to characterize longitudinal salivary RNA expression in 600 children with mTBI and identify RNA patterns that predict length and characterof concussive symptoms, as well as the response to therapy.

Hypothesis: Specific RNAs will be differentially regulated in children with prolonged mTBI symptoms across the acute and sub-acute time periods. The investigators predict that a set of RNAs with differential expression in children with mTBI will be statistically associated with functional measures of mTBI symptoms as well as the duration of concussive symptoms.

Rationale: Preliminary studies show that miRNA is altered in adults with varying degrees of TBI and that salivary RNA is altered by disorders of the CNS. These studies indicate that serum-based miRNA may be used as an accurate biomarker for differentiating adults with and without TBI. Whether similar patterns can seen in the saliva of children following mTBI remains to be seen. Furthermore, the influence of confounding variables such as gender, mechanism of injury, and previous mTBIs on RNA profiles has not been explored. The investigators propose to investigate these questions by examining salivary RNA from 600 children (ages five to twenty-one years) with a clinical diagnosis of mTBI (as well as 100 age-and gender-matched controls, recruited from the Penn State Pediatric Concussion Clinic, Emergency Department, and the affiliated primary care clinics). The investigators plan to prospectively follow 600 children with mTBI for 1-month post-concussion, tracking subjective symptoms with the Child Sports Concussion Assessment Tool (SCAT-5), and objective symptoms of balance and cognition. Saliva will be collected via swab at three time-points (at initial clinical presentation, 1-2 weeks, and 4-weeks after the date of initial mTBI). Expression of salivary RNA taken at initial presentation will be compared against symptom duration (where prolonged post-concussive symptoms are defined as those lasting >4 weeks) and character (as measured numerically by Post-concussion symptom inventory self-report and ClearEdge scoring). The investigators plan to identify a set of salivary RNAs that can easily be used to predict clinical course for pediatric patients following a diagnosis of mTBI.

ELIGIBILITY:
Inclusion Criteria:

* 5-21 years with mild traumatic brain injury that occurred within 7 days of enrollment

Exclusion Criteria:

* Sever traumatic brain injury
* Skull fracture
* Concurrent upper respiratory infection
* Patients whose primary language is not English
* Periodontal infection
* Wards of the state
* Ongoing seizure disorder,
* Drug or alcohol dependency

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children 5-21 years with mild traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of concussion symptoms | 4-weeks post injury
  subjective (score >7 on PCSI) or objective (score outside 85 percentile on accelerometer balance testing or cognitive testing)

SECONDARY OUTCOMES:
Salivary RNA profile | Within 7d of initial injury, 1-2 weeks post-injury, and 4-weeks post-injury
  measured with RNAseq

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hicks, MD, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No